CLINICAL TRIAL: NCT07063966
Title: Are Developmentally At Risky Babies Environmentally Disadvantaged?
Status: Not yet recruiting | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Seda AYAZ TAŞ, Assistant Professor, Abant Izzet Baysal University
Other Study IDs: BAIBU-FTR-SAT-12
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Risky Baby; Motor Development; Sensory Profiles; Environmental Conditions
Keywords: risky baby; motor development; sensory profiles; environmental conditions

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- risky babies: High-risk infants are defined as those exposed to adverse biological or environmental factors that increase the risk of neurodevelopmental issues. Prenatal risk factors include maternal substance use, chronic illnesses, infections, and complications such as intrauterine growth restriction or multiple pregnancies. Natal risks involve preterm or postterm birth, birth trauma, and perinatal asphyxia. Postnatal risks include low or high birth weight, neonatal infections, respiratory problems, and feeding difficulties. Additionally, infants with genetic conditions like Down syndrome, epilepsy, or neuromuscular diseases are considered developmentally at risk.
- control group: Typically developing children were included as the control group to provide a comparative baseline for assessing developmental differences.

SUMMARY:
A study conducted on infants aged between 3 and 11 months revealed a positive relationship between the home environment and developmental outcomes. Similarly, another study found that variability in motor and cognitive development could be better explained by environmental factors and parental knowledge and practices. It has also been shown that the opportunities provided in the home environment of preterm infants may be associated with motor development and sensory processing skills. In the literature, it is generally observed that studies evaluate either term infants or both preterm and term infants together. In the present study, however, infants at developmental risk and typically developing infants will be evaluated separately.

The aim of this study is to assess whether infants at developmental risk are disadvantaged in terms of their home environment.

The hypotheses of this study are as follows:

H1-1: There is a difference in environmental arrangements between typically developing infants and those at developmental risk.

H1-2: There is a relationship between home environmental arrangements and motor development.

H1-3: There is a relationship between home environmental arrangements and sensory profile.

DETAILED DESCRIPTION:
A "high-risk infant" is defined as a baby who has experienced any adverse environmental or biological factors in their medical history and is therefore at increased risk for neurodevelopmental problems. Exposure to various factors during the prenatal, natal, and postnatal periods may negatively affect the development of these infants.

In the prenatal period, maternal use of medications, alcohol, or tobacco; chronic maternal illnesses (such as diabetes, hypertension, congenital heart disease, or renal failure); infections during pregnancy; congenital anomalies; intrauterine growth restriction; multiple pregnancies; preeclampsia; eclampsia; and placenta previa are considered risk factors for the baby. During the natal period, complications such as preterm or postterm birth, premature rupture of membranes, birth trauma, perinatal asphyxia, intrauterine hemorrhage, and meconium aspiration may threaten infant health. In the postnatal period, birth weight below 2500 grams or above 4000 grams, neonatal sepsis and meningitis, intraventricular hemorrhage, feeding difficulties, hypoglycemia, respiratory distress syndrome, respiratory failure, a history of ventilator support, and hyperbilirubinemia are considered developmental risk factors.

Infants diagnosed with Down syndrome, rare genetic disorders, epilepsy/seizure disorders, or neuromuscular diseases are also classified as developmentally at-risk. Due to these diverse factors, infants at risk may not develop typically. These infants are vulnerable to developmental delays and neurodevelopmental disorders that may affect motor skills, cognitive abilities, and sensory processing. High-risk infants, such as those born prematurely, often demonstrate impairments in both gross and fine motor skills. It has been reported that individuals born very preterm and with very low birth weight, but without cerebral palsy, still exhibit significant motor impairments compared to their term-born peers.

Preterm infants are also at increased risk for difficulties in social-emotional, cognitive, language, and sensory processing domains. It has been shown that infants born before 32 weeks of gestation often experience challenges in sensory processing. In one study, preterm infants demonstrated altered sensory processing patterns, with reduced responses to deep tactile pressure and vestibular input. A positive association has been observed between motor development and sensory processing, and delayed gross motor development is more likely in preterm infants who display abnormal sensory processing and poor postural control. These developmental limitations can worsen as the child grows, especially in environments lacking sufficient developmental stimulation.

Environmental factors encompass the physical, social, and behavioral settings in which an individual lives. A rich and stimulating environment during early life has been shown to support stronger neural connections in the brain and contribute positively to a child's overall development-including motor, language, cognitive, and literacy skills. During the first years of life, children spend most of their time in the home environment. Therefore, the home plays a critical role in early childhood development, and the presence of various stimulating materials during this period is of great importance. A supportive home environment includes educational materials such as toys and books, adequate physical space, and stimuli provided by family members. Research has shown that family support, environmental conditions, and interactions with toys positively influence children's motor, social, and cognitive development. During infancy and early childhood, sensory processing enables learning by integrating experiences and forms the foundation for more advanced perceptual and cognitive abilities. In this context, motor development and sensory processing are complementary and mutually supportive developmental processes.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria (Developmentally At-Risk Infants):

Infants classified as developmentally at risk

Aged between 7 and 18 months

Parental consent for participation in the study

Inclusion Criteria (Typically Developing Infants):

Aged between 7 and 18 months

Parental consent for participation in the study

Exclusion Criteria:

* Infants with unstable vital signs

Infants currently hospitalized

Ages: 7 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants who were developmentally at risk, aged between 7 and 18 months, and whose parents consented voluntarily were included in the study. Infants who were hospitalized or had unstable vital signs were excluded. Typically developing infants aged 7 to 18 months with parental consent were included as the control group. Written informed consent was obtained from the parents of all participating infants.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2025-07-03 (Estimated); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-11-10 (Estimated)

PRIMARY OUTCOMES:
Assessment of Home Environment Supporting Motor Development - Infant Scale (AHEMD-IS): | 2 year
  The AHEMD-SR, developed in 2005, evaluates the home environment of children aged 18-42 months. Recently, the 3-18 month version (AHEMD-IS) was validated to assess the quality and quantity of motor development opportunities at home. The scale has 41 items across four domains: Physical Space (indoor/outdoor), Variety of Stimulation, Gross Motor Toys, and Fine Motor Toys. Home environments are rated as excellent, adequate, moderate, or inadequate. For infants 3-11 months, 32 items are applicable; 12-18 months respond to all items. Responses include yes/no (0/1) and frequency scales from never (0) to always (3). Maximum scores are 66 for under 12 months and 93 for older infants; higher scores indicate better environmental enrichment. Turkish validity and reliability were confirmed with Cronbach's alpha of 0.846 and ICC of 0.830. Author permission was obtained.

SECONDARY OUTCOMES:
Alberta Infant Motor Scale (AIMS): | 2 year
  AIMS is a standardized tool assessing gross motor development from birth to independent walking (up to 18 months). It identifies motor delays, monitors progress pre- and post-intervention, and evaluates rehabilitation effectiveness. Infants are observed in four positions: prone, supine, sitting, and standing. Movements related to weight-bearing, posture, and antigravity are scored. Each observed movement scores 1, unobserved 0, focusing on the "developmental window" of the two most mature movements. Scores per position are summed for a raw score, converted to age-based percentiles to assess motor level. Assessment takes 20-30 minutes, ideally with caregiver present for infant comfort. AIMS is widely used to profile infant motor development.
Sensory Profile Assessment: | 2 year
  The Toddler Sensory Profile-2 (7-35 months) is a parent-report questionnaire designed to evaluate sensory processing in infants. It consists of 54 items and takes approximately 15 minutes to complete. In this study, it will be applied to infants aged 7-18 months. Parents rate the frequency of their child's responses to various sensory experiences on a 5-point scale: Almost Always (5), Often (4), Sometimes (3), Rarely (2), Almost Never (1), with an additional "Not Applicable" option. Total raw scores are classified using normative curves and sensory classification as follows: (i) Much less than others (<2%), (ii) Less than others (1-2 SD below mean), (iii) Similar to most (±1 SD), (iv) More than others (1-2 SD above mean), (v) Much more than others (>98%).
Bayley Scales of Infant and Toddler Development - Third Edition (Bayley-III): | 2 year
  Bayley-III is a reliable and valid tool for assessing cognitive, language, and motor development in children aged 0-42 months. It identifies developmental delays and aids intervention planning. The scale provides raw scores, standard scores, percentile ranks, and growth scores, detailing performance in subscales: Cognitive, Receptive and Expressive Communication, Fine Motor, and Gross Motor. Scoring awards 1 point for correct and 0 for incorrect responses. Developmental scores range from 200 to 800 (mean=500, SD=100). The test follows basal and ceiling rules for item administration. Assessment requires a quiet, well-lit environment, fostering a warm, trusting interaction. Materials are engaging and hygienically maintained. Bayley-III is widely used by multidisciplinary teams for diagnosis and research, especially in early intervention. The research team's certified examiner will conduct the assessment.

CONTACTS AND LOCATIONS:
Locations (3):
- Turkey (Türkiye) (3):
  - Kdz. Ereğli Gökkuşağı Özel Eğitim ve Rehabilitasyon Merkezi, Zonguldak, Ereğli
  - Bolu Abant İzzet Baysal University, Bolu
  - Düzce Gökkuşağı Özel Eğitim ve Rehabilitasyon Merkezi, Düzce

IPD SHARING:
Plan to Share IPD: No